CLINICAL TRIAL: NCT06134635
Title: Short-term Effect of Proprotein Convertase Subtilisin/Kexin Type 9 Inhibitor in Chinese Population With Acute Ischemic Stroke: the Singe-center Real-world Study
Brief Title: Short-term Effect of PCSK9 Inhibitor in Patients With Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: RMeng
Record Dates: First submitted 2023-10-24; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Evolocumab; PCSK9 Inhibitor; Statins
MeSH Terms: conditions — Ischemic Stroke | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; evolocumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Statin-alone group: The participants in statin-alone group receive statins alone for lipid reduction.
  Interventions: Drug: Statins
- PCSK9-i group: The participants in PCSK9-i group receive statins and evolocumab for lipid reduction.
  Interventions: Drug: Statins; Drug: Evolocumab

INTERVENTIONS:
Drug: Statins — Atorvastatin 20mg qn or rosuvastatin 10mg qn or pivastatin 2mg qn, oral
  Other Names: statin therapy
Drug: Evolocumab — Evolocumab 140mg twice a month, subcutaneous injection
  Other Names: PCSK9-i
  Groups: PCSK9-i group

SUMMARY:
This is a prospective cohort study to investigate the early impact of evolocumab on patients with acute ischemic stroke (AIS) in China. Evolocumab, a proprotein convertase subtilisin/kexin taye 9 inhibitor, can significantly reduce low density lipoprotein cholesterol (LDL-C) levels and has a positive effect on improving cardiovascular events. However, existing studies have focused almost exclusively on the long-term effects of Evolocumab, and the early effects of Evolocumab on AIS patients remains unclear.

DETAILED DESCRIPTION:
Patients aged 18-80 years old admitted to the Department of Neurology, Xuanwu Hospital, Capital Medical University, with a definite diagnosis of acute ischemic stroke and receiving lipid-lowering therapy with statins with or without evolocumab will be included in this study. Participants will be divided into two groups according to the lipid-lowering therapy they used: 1) statin-alone group: the participants receive statins alone (atorvastatin 20mg qn or rosuvastatin 10mg qn or pivastatin 2mg qn) for lipid reduction, and 2) PCSK9-i group: the participants receive statins (atorvastatin 20mg qn or rosuvastatin 10mg qn or pivastatin 2mg qn) and evolocumab (140mg twice a month) for lipid reduction. Most importantly, the lipid-lowering therapy of participants will be decided only by clinicians not involved in the study, not by the investigators. The levels of blood lipid (TC, TG, HDL-C, LDL-C, Apo AI and Apo B) and inflammatory biomarkers (hsCRP and IL-6) of these participants at different time points (day 1, day 3, day 5, and month 3) will be recorded. The target level of LDL-C is the LDL-C reduction ≥50% from the baseline and LDL-C<1.4mmol/L (55mg/dL). In addition, the cardiovascular events and adverse drug reactions of these participants during follow-up will also be recorded. During the follow-up period (3 months), participants who changed their lipid-lowering regimen, including the type, dosage and frequency of statins and evolocumab, will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute ischemic stroke;
* Aged 18-80 years, gender unlimited;
* The fasting LDL-C≥1.8mmol/L (70mg/dL);
* Received lipid-lowering therapy with statins with or without evolocumab;
* Premorbid mRS ≤ 2;
* NIHSS ≤ 15;
* Subjects participated in the study voluntarily and signed informed consent.

Exclusion Criteria:

* Participants who changed their lipid-lowering regimen;
* Participants allergic to PCSK9 inhibitors;
* Participants treated with cholesterol ester transfer protein inhibitor within 12 months prior to enrollment;
* LDL or plasma apheresis within 12 months prior to enrollment；
* Last known left ventricular ejection fraction < 30%
* Known hemorrhagic stroke at any time；
* Severe renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) < 20 mL/min/1.73m2 at final screening；
* Active liver disease or hepatic dysfunction, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times；
* Pregnant or lactating women；
* Severe, concomitant non-cardiovascular disease that is expected to reduce life expectancy to less than 3 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients aged 18 to 80 years
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
LDL-C target achievement rate on Day 5, Month 3 | Day 5, Month 3
  LDL-C target achievement rate= Number of patients who achieved the LDL-C target level/ Total number of follow-up patients

SECONDARY OUTCOMES:
Percentage change in LDL-C level on Day 1, Day 3, Day 5, and Month 3 | Day 1, Day 3, Day 5, Month 3
  Percentage change in LDL-C level= (follow-up LDL-C level - baseline LDL-C level)/ baseline LDL-C level
Percentage change in HDL-C level on Day 1, Day 3, Day 5, and Month 3 | Day 1, Day 3, Day 5, Month 3
  Percentage change in HDL-C level= (follow-up HDL-C level - baseline HDL-C level)/ baseline HDL-C level
Percentage change in TC level on Day 1, Day 3, Day 5, and Month 3 | Day 1, Day 3, Day 5, Month 3
  Percentage change in TC level= (follow-up TC level - baseline TC level)/ baseline TC level
Percentage change in TG level on Day 1, Day 3, Day 5, and Month 3 | Day 1, Day 3, Day 5, Month 3
  Percentage change in TG level= (follow-up TG level - baseline TG level)/ baseline TG level
Percentage change in Apo AI level on Day 1, Day 3, Day 5, and Month 3 | Day 1, Day 3, Day 5, Month 3
  Percentage change in Apo AI level= (follow-up Apo AI level - baseline Apo AI level)/ baseline Apo AI level
Percentage change in Apo B level on Day 1, Day 3, Day 5, and Month 3 | Day 1, Day 3, Day 5, Month 3
  Percentage change in Apo B level= (follow-up Apo B level - baseline Apo B level)/ baseline Apo B level
Percentage change in hsCRP level on Day 1, Day 3, Day 5, and Month 3 | Day 1, Day 3, Day 5, Month 3
  Percentage change in hsCRP level= (follow-up hsCRP level - baseline hsCRP level)/ baseline hsCRP level
Percentage change in IL-6 level on Day 1, Day 3, Day 5, and Month 3 | Day 1, Day 3, Day 5, Month 3
  Percentage change in IL-6 level= (follow-up IL-6 level - baseline IL-6 level)/ baseline IL-6 level
Percentage of mRS≤2 on Month 3 | Month 3
  Percentage of mRS≤2= Number of patients with mRS≤2/ Total number of follow-up patients
Incidence of major cardiovascular events on Month 3 | Month 3
  Major cardiovascular events: stroke, cardiovascular death, myocardial infarction, hospitalization for unstable angina, and coronary revascularization.
Incidence of adverse events on Month 3 | Month 3
  Adverse events: injection site reaction, anaphylaxis, myopathy, abnormal liver function, new onset diabetes, cognitive impairment, and hemorrhagic cerebral infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Ran, PhD, Study Chair — Xuanwu Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No